CLINICAL TRIAL: NCT00254371
Title: Pathogenesis of Sarcopenia and Metabolic Changes in Aging
Brief Title: DHEA and Testosterone Replacement in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 547-96; P01AG014383 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Aging; Low DHEA for Women; Low Testosterone and DHEA for Men

INTERVENTIONS:
Procedure: Androgen Replacement

SUMMARY:
Sarcopenia is a major health problem among the rapidly expanding elderly population in our society. Disabilities directly related to muscle weakness, and indirectly related to changes in body composition and metabolic dysfunctions, are causing a staggering toll in disability and health care costs.

Osteopenia occurs almost simultaneously with sarcopenia in the elderly population and muscle weakness increases the risk for falls and therefore, fractures. Although these issues have been separate addressed in several studies, an integrated investigational approach to better understand the pathogenesis of sarcopenia and other age-related metabolic abnormalities and to investigate the potential role of androgens have not been undertaken in a comprehensive manner.

The program contains four independent research programs, each representing different research disciplines, and four separate cores supporting the four projects.

The main focus of the project is to determine the effect of the replacement of testosterone in elderly men and DHEA in elderly men and women and to compare these effects with placebo treatment over a two-year period.

Project 1, "Effect of Androgen Replacement on Muscle Metabolism" will specifically determine whether these interventions have a differential effect on size and quality of muscle in terms of strength and metabolic functions. Project 2, "Effect of Androgen Replacement on Bone Metabolism," will determine the effects of this intervention on bone mineral density and markers of bone turnover.

Project 3, "The Effect of Androgen Replacement on Carbohydrate Metabolism," will determine whether the age-associated decrease in circulating androgens contributes to the alterations in carbohydrate metabolism that are commonly observed in the elderly and on insulin action, insulin secretion, and glucose effectiveness.

Project 4, "Effect of Androgen Replacement on Fat Metabolism" will determine whether changes in fat distribution that occur with aging could result from differences in regional fatty acid uptake and systemic fatty acid kinetics, and whether these determinants of fat distribution are altered by the interventions.

The data emerging from these studies will be integrated to determine the intervention of sarcopenia with other metabolic changes and hopefully will contribute to a better understanding of muscle, bone, carbohydrate and fat metabolism.

This study will hopefully form the scientific basis for future trials of androgen replacement in the elderly.

ELIGIBILITY:
Inclusion criteria:

bioavailable testosterone less than 103 nanogram/dl and DHEA-S level less than 157 microgram/dl for men; DHEA-S less than 95 microgram/dl for women;

Exclusion criteria:

significant ischemic heart disease, renal disease, uncontrolled hypertension, diabetes mellitus, malignancy, malabsorption, bone disorders, chronic obstructive pulmonary disease, or sleep apnea.

Others exclusion criteria include abnormal serum calcium, phosphorus, alkaline phosphatase, asparate aminotransferase, creatinine, urinary calcium, thyroid stimulating hormone, and erythrocyte sedimentation rate.

People taking medication that may affect outcome measures such as adrenal steroids, anticonvulsant therapy thiazide diuretics, and estrogen replacement were also excluded. People engaged in a regular exercise program lasting more than 20 minutes more than two times per week and those men whose PSA level (age adjusted upper limit) were also excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1998-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
physical performance (VO2 peak, muscle strength as measured by chest press, double knee extension, and isokinetic knee extension
body composition (fat percent, fat free mass, abdominal visceral fat, and thigh muscle area)
bone parameters (BMD of ultradistal radius, femur neck, femur total and anterior-posterior of L2-L4 spine
fasting plasma insulin and glucose

SECONDARY OUTCOMES:
quality of life
glucose and insulin after mixed meal
muscle protein synthesis
hormone levels
prostate size

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Nair KS, Rizza RA, O'Brien P, Dhatariya K, Short KR, Nehra A, Vittone JL, Klee GG, Basu A, Basu R, Cobelli C, Toffolo G, Dalla Man C, Tindall DJ, Melton LJ 3rd, Smith GE, Khosla S, Jensen MD. DHEA in elderly women and DHEA or testosterone in elderly men. N Engl J Med. 2006 Oct 19;355(16):1647-59. doi: 10.1056/NEJMoa054629. PMID 17050889
- [Derived] Gonzalez Lopez JS, Nielsen S, Jensen MD. Meal fatty acid metabolism is associated with long-term weight gain in women - a retrospective cohort study. Am J Clin Nutr. 2026 Jan 28:101219. doi: 10.1016/j.ajcnut.2026.101219. Online ahead of print. PMID 41617091
- [Derived] Espinosa De Ycaza AE, Rizza RA, Nair KS, Jensen MD. Effect of Dehydroepiandrosterone and Testosterone Supplementation on Systemic Lipolysis. J Clin Endocrinol Metab. 2016 Apr;101(4):1719-28. doi: 10.1210/jc.2015-4062. Epub 2016 Feb 17. PMID 26885881
- [Derived] Bush NC, Basu R, Rizza RA, Nair KS, Khosla S, Jensen MD. Insulin-mediated FFA suppression is associated with triglyceridemia and insulin sensitivity independent of adiposity. J Clin Endocrinol Metab. 2012 Nov;97(11):4130-8. doi: 10.1210/jc.2012-2285. Epub 2012 Aug 29. PMID 22933539
- [Derived] Srinivasan M, Irving BA, Frye RL, O'Brien P, Hartman SJ, McConnell JP, Nair KS. Effects on lipoprotein particles of long-term dehydroepiandrosterone in elderly men and women and testosterone in elderly men. J Clin Endocrinol Metab. 2010 Apr;95(4):1617-25. doi: 10.1210/jc.2009-2000. Epub 2010 Feb 5. PMID 20139233